CLINICAL TRIAL: NCT03862807
Title: An Open-label Study to Evaluate Safety, Efficacy and Pharmacokinetics (PK) of Patisiran-LNP in Patients With Hereditary Transthyretin-mediated Amyloidosis (hATTR Amyloidosis) With Disease Progression Post-Orthotopic Liver Transplant
Brief Title: Patisiran in Patients With Hereditary Transthyretin-mediated Amyloidosis (hATTR Amyloidosis) Disease Progression Post-Liver Transplant
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALN-TTR02-008; 2018-003519-24 (EudraCT Number)
Record Dates: First submitted 2019-02-28; First posted 2019-03-05 (Actual); Results first posted 2021-12-21 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2021-11

CONDITIONS: Amyloidosis, Familial; Transthyretin Amyloidosis
MeSH Terms: conditions — Amyloidosis, Familial; Amyloidosis, Hereditary, Transthyretin-Related | interventions — patisiran

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Patisiran (Experimental): Participants received patisiran 0.3 milligrams/kilogram (mg/kg) via intravenous (IV) infusion once every 3 weeks (q3w) for 12 months. Dosing was based on actual body weight. For participants weighing 100 kg or more, patisiran was administered at a total dose of 30 mg IV q3w.
  Interventions: Drug: Patisiran

INTERVENTIONS:
Drug: Patisiran — Patisiran was administered via IV infusion.
  Other Names: ALN-TTR02; ONPATTRO

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and pharmacokinetics of patisiran in participants with hereditary transthyretin-mediated amyloidosis (hATTR amyloidosis) with disease progression after liver transplant.

ELIGIBILITY:
Inclusion Criteria:

* Received liver transplant for treatment of hATTR amyloidosis ≥12 months before study start
* Has increase in polyneuropathy disability (PND) score after liver transplant
* Has received stable immunosuppressive regimen with ≤10 mg/day of prednisone for at least 3 months before study start
* Has Karnofsky Performance Status (KPS) of ≥70%
* Has vitamin A level greater than or equal to lower limit of normal

Exclusion Criteria:

* Has previously received inotersen or patisiran
* Has clinically significant liver function test abnormalities
* Has known portal hypertension with ascites
* Has estimated glomerular filtration rate (eGFR) ≤30 mL/min/1.73 m^2
* Has known leptomeningeal amyloidosis
* Has infection with hepatitis B, hepatitis C or human immunodeficiency virus (HIV)
* Has New York Heart Association heart failure classification of >2
* Is wheelchair bound or bedridden
* Has received organ transplants other than liver transplant
* Will be using another tetramer stabilizer during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2020-10-06 (Actual); Study Completion 2020-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals
Locations (9):
- France (2):
  - Clinical Trial Site, Créteil
  - Clinical Trial Site, Le Kremlin-Bicêtre
- Clinical Trial Site, Münster, Germany
- Clinical Trial Site, Messina, Italy
- Clinical Trial Site, Porto, Portugal
- Spain (2):
  - Clinical Trial Site, Barcelona
  - Clinical Trial Site, Huelva
- Clinical Trial Site, Umeå, Sweden
- Clinical Trial Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Access to Anonymized individual participant data that support these results is made available 12 months after study completion and not less than 12 months after the product and indication have been approved in the US and/or the EU.
  Data will be provided contingent upon the approval of a research proposal and the execution of a data sharing agreement. Requests for access to data can be submitted via the website www.vivli.org.

REFERENCES:
- [Derived] Badri P, Habtemariam B, Melch M, Clausen VA, Arum S, Li X, Jay PY, Vest J, Robbie GJ. Pharmacokinetics and Pharmacodynamics of Patisiran in Patients with hATTR Amyloidosis and with Polyneuropathy After Liver Transplantation. Clin Pharmacokinet. 2023 Oct;62(10):1509-1522. doi: 10.1007/s40262-023-01292-w. Epub 2023 Aug 28. PMID 37639169
- [Derived] Schmidt HH, Wixner J, Plante-Bordeneuve V, Munoz-Beamud F, Llado L, Gillmore JD, Mazzeo A, Li X, Arum S, Jay PY, Adams D; Patisiran Post-LT Study Group. Patisiran treatment in patients with hereditary transthyretin-mediated amyloidosis with polyneuropathy after liver transplantation. Am J Transplant. 2022 Jun;22(6):1646-1657. doi: 10.1111/ajt.17009. Epub 2022 Mar 26. PMID 35213769
- [Derived] Seibert K, Wlodarski R, Sarswat N, Appelbaum D, Issa NP, Soliven B, Rezania K. Progressive Multiple Mononeuropathy in a Patient With Familial Transthyretin Amyloidosis After Liver Transplantation. J Clin Neuromuscul Dis. 2022 Mar 1;23(3):143-147. doi: 10.1097/CND.0000000000000368. PMID 35188911

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with hereditary transthyretin-mediated amyloidosis (hATTR amyloidosis) with disease progression post-orthotopic liver transplant were enrolled at nine sites in France, Germany, Italy, Portugal, Spain, Sweden and the United Kingdom.
Period: Overall Study
Arm/Group | Patisiran
Started | 24
Treated | 23
Completed Treatment | 22
Completed | 23
Not Completed | 1
Not completed — Not Treated Due to Eligibility Criteria Failure | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All participants who received any amount of patisiran.
Arm/Group | Patisiran
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 22
  Asian | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 23
Serum Transthyretin (TTR) [Median (Full Range); unit: mg/L] | 192.140 [123.74 to 315.12]

OUTCOME MEASURES:

1. Primary Outcome: Average of Month 6 and Month 12 Percentage Reduction From Baseline in Serum Transthyretin (TTR)
Description: Serum TTR was assessed using enzyme linked immunosorbent assay (ELISA). The average of the percentage reduction in serum TTR observed at Month 6 and at Month 12 is first calculated for each patient and then the median (95% CI) of these averaged values is summarized for the Safety Analysis Set.
Time Frame: Baseline, Months 6 and 12
Population: Safety Analysis Set: All participants who received any amount of patisiran.
Measure: Median (95% Confidence Interval); unit: percent reduction
Arm/Group | Patisiran
Number analyzed (Participants) | 22
percent reduction | 91.0 [86.1 to 92.3]

2. Secondary Outcome: Change From Baseline in the Neuropathy Impairment Score (NIS) at Month 12
Description: The NIS is a composite neurologic impairment score that assesses motor weakness (NIS-W), sensation (NIS-S) and reflexes (NIS-R) by physical exam. The minimum and maximum values are 0 and 244, respectively. A higher score indicates a worse outcome.
Time Frame: Baseline, Month 12
Population: Participants from the Per Protocol (PP) Analysis Set, all participants in the Safety Analysis Set who missed ≤2 doses of patisiran due to the COVID-19 pandemic during the study, with NIS data available at Month 12.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Patisiran
Number analyzed (Participants) | 20
score on a scale | -3.7 (2.7)

3. Secondary Outcome: Change From Baseline in Norfolk Quality of Life-Diabetic Neuropathy (Norfolk QoL-DN) Score at Month 12
Description: The Norfolk QoL-DN questionnaire is a standardized 35-item patient-reported outcomes measure that is sensitive to the different features of diabetic neuropathy - small fiber, large fiber, and autonomic nerve function. The minimum and maximum values are -4 and 136, respectively. A higher score indicates a worse outcome.
Time Frame: Baseline, Month 12
Population: Per Protocol (PP) Analysis Set: All participants in the Safety Analysis Set who missed ≤2 doses of patisiran due to the COVID-19 pandemic during the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Patisiran
Number analyzed (Participants) | 21
score on a scale | -6.5 (4.9)

4. Secondary Outcome: Change From Baseline in the Rasch-Built Overall Disability Scale (R-ODS) at Month 12
Description: The R-ODS is comprised of a 24-item linearly weighted scale that specifically captures activity and social participation limitations. The minimum and maximum values are 0 and 48, respectively. A higher score indicates a better outcome.
Time Frame: Baseline, Month 12
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Patisiran
Number analyzed (Participants) | 21
score on a scale | -0.1 (1.1)

5. Secondary Outcome: Change From Baseline in the Composite Autonomic Symptom Score (COMPASS-31) at Month 12
Description: The COMPASS-31 questionnaire is a measure of autonomic neuropathy symptoms. The questions evaluate 6 autonomic domains (orthostatic intolerance, vasomotor, secretomotor, gastrointestinal, bladder, and pupillomotor). The minimum and maximum values are 0 and 100, respectively. A higher score indicates a worse outcome.
Time Frame: Baseline, Month 12
Population: Participants from the Per Protocol (PP) Analysis Set, all participants in the Safety Analysis Set who missed ≤2 doses of patisiran due to the COVID-19 pandemic during the study, with COMPASS-31 data available at Month 12.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Patisiran
Number analyzed (Participants) | 20
score on a scale | -5.0 (2.6)

6. Secondary Outcome: Change From Baseline in the Modified Body Mass Index (mBMI) at Month 12
Description: Nutritional status of participants was evaluated using the mBMI, calculated as BMI (kg/m^2) multiplied by albumin (g/L). An increase from baseline in mBMI suggests improvement, and a decrease from baseline suggests worsening.
Time Frame: Baseline, Month 12
Population: as for outcome 3
Measure: Mean (Standard Error); unit: (kg/m^2)*(g/L)
Arm/Group | Patisiran
Number analyzed (Participants) | 21
(kg/m^2)*(g/L) | 4.4 (21.8)

7. Secondary Outcome: Percentage of Participants With Adverse Events
Description: An AE is any untoward medical occurrence in a participant or clinical investigational patient administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Time Frame: From baseline to end of study at Month 13
Population: Safety Analysis Set: All participants who received any amount of patisiran.
Measure: Number; unit: percentage of participants
Arm/Group | Patisiran
Number analyzed (Participants) | 23
percentage of participants | 100

ADVERSE EVENTS:
Time Frame: From baseline to end of study at Month 13.
Description: Safety Analysis Set: All participants who received any amount of patisiran.
Arm/Group | Patisiran
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 5/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patisiran (N=23)
Atrial thrombosis (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 3
Cholangitis (Hepatobiliary disorders) | 1
Infusion related reaction (Immune system disorders) | 1
Pneumonia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Syncope (Nervous system disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Patisiran (N=23)
Vertigo (Ear and labyrinth disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Bile acid malabsorption (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 8
Asthenia (General disorders) | 2
Chest pain (General disorders) | 2
Fatigue (General disorders) | 3
Oedema peripheral (General disorders) | 5
Pyrexia (General disorders) | 3
Infusion related reaction (Immune system disorders) | 6
Bronchitis (Infections and infestations) | 2
Cystitis (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 3
Skin laceration (Injury, poisoning and procedural complications) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5
Headache (Nervous system disorders) | 3
Oliguria (Renal and urinary disorders) | 2
Poor venous access (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
It is intended that after completion of the study, the data are to be submitted for publication in a scientific journal and/or for reporting at a scientific meeting. A separate publication by Institution or PI may not be submitted for publication until after this primary manuscript is published or following 12 months after completion of the study. A copy of any proposed publication based on this study, must be provided and confirmed received at the Sponsor at least 30 days before its submission.

DOCUMENTS (2):
  • Study Protocol (2018-10-07): https://cdn.clinicaltrials.gov/large-docs/07/NCT03862807/Prot_002.pdf
  • Statistical Analysis Plan (2020-10-08): https://cdn.clinicaltrials.gov/large-docs/07/NCT03862807/SAP_003.pdf